CLINICAL TRIAL: NCT01856010
Title: Short-term Efficacy and Cognitive Side Effects of Acute Electroconvulsive Therapy (ECT) for Agitation and Aggression in Dementia
Brief Title: Study of Electroconvulsive Therapy (ECT) Treatment for Agitation and Aggression in Dementia
Status: Completed | Type: Observational
Sponsor: Pine Rest Christian Mental Health Services (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SM10-1221-01
Record Dates: First submitted 2012-11-13; First posted 2013-05-17 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Dementia; Aggression; Agitation
Keywords: Dementia; Aggression; Agitation
MeSH Terms: conditions — Dementia; Aggression; Psychomotor Agitation | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ECT Treatment: Those who were referred for ECT treatment for behavior refractory to standard care and who opted to undergo ECT treatment
  Interventions: Other: ECT treatment
- Standard Care (Non-ECT Group): Those who were referred for ECT treatment for behavior refractory to standard care, but who opted to not undergo ECT treatment and continue with standard care.
  Interventions: Other: Standard Care (Non-ECT group)

INTERVENTIONS:
Other: ECT treatment — The decision to administer ECT treatment will have already been made before the subject is approached about study participation. Only individuals who were referred for ECT due to behavior refractory to standard care will be eligible to participate. If they decide to do ECT treatment, they are in the ECT group.
  Groups: ECT Treatment
Other: Standard Care (Non-ECT group) — The decision to administer ECT treatment will have already been made before the subject is approached about study participation. Only individuals who were referred for ECT due to behavior refractory to standard care will be eligible to participate. If they decide not to do ECT treatment and continue with standard care, they are in the Standard Care (Non-ECT) Group.
  Groups: Standard Care (Non-ECT Group)

SUMMARY:
Agitation/aggression is one of the most common and serious behavioral complications of dementia. If the behavior is refractory to standard care (behavior approaches and off label use of psychotropic medications), other evidence based treatment options are not currently available. Retrospective reviews and preliminary studies have indicated Electroconvulsive Therapy (ECT) may be a safe, effective intervention in this patient population. This study will measure the impact of open-label ECT on symptoms of agitation, aggression, cognition, mood and psychosis for patients referred for ECT who accept this intervention vs. those patients referred for ECT but decline this intervention (i.e. standard care controls). It will also assess adverse events, activities of daily living and caregiver burden during study participation. The hypothesis is that subjects with dementia related aggression/agitation who receive ECT will show significantly greater reductions in these behaviors than subjects who do not consent for ECT and continue with standard care. Pine Rest is partnering with McLean Hospital (Massachusetts) to answer this question. To our knowledge, this is the first prospective study to examine whether patients receiving ECT or standard care differ in reduction of aggression and agitation symptom severity and changes in cognition pre- and post- treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 50 years or older from the Older Adult Unit of Pine Rest Christian Mental Health Services or Geriatric Unit at McLean Hospital
* Diagnosis of Dementia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) Criteria
* Mini Mental Status Examination (MMSE) score of 16 or greater
* Fluent in English
* Presence of agitation/aggression symptoms as defined by a minimum aggression score on the Cohen-Mansfield Agitation Inventory Short Version (CMAI): a score of 4 or greater on at least one aggressive item, or a score of 3 on at least 2 aggressive items, or a score of 2 on at least 3 aggressive items, or 2 aggressive items occuring in frequency of 2 and 1 at frequency of 3.
* A therapeutic decision will have already been made by the treating psychiatrist in consultation with the ECT team to use ECT treatment for agitation and aggression associated with dementia, with or without depression/mania. Patients will be included in the ECT treatment group if their legal representative consents to ECT treatment. Patients whose legal representative does not consent to ECT treatment will be included in the Standard Care (Non-ECT) treatment group.
* Informed Consent signed by authorized legal guardian and assent given by the participant
* Signed Authorization for Release of Healthcare Information by authorized legal guardian

Exclusion Criteria:

* Current diagnosis of co-morbid delirium according to DSM-IV upon study entry
* ECT treatment within 90 days prior to study enrollment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals age 50 or older that have been diagnosed with dementia and associated agitation and aggression and have already been referred for ECT.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in baseline of the Cohen-Mansfield Agitation Inventory Short Version (CMAI) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Measures agitation or aggression outcomes - completed by primary caregiver

SECONDARY OUTCOMES:
Severe Impairment Battery (SIB) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Gathers direct performance-based data from the subject with dementia on a wide variety of low-level tasks that take into account the specific behavioral and cognitive deficits associated with severe dementia
Cornell Scale for Depression in Dementia (CSDD) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Assesses the presence and severity of depressive symptoms - completed by primary caregiver
Neuropsychiatric Inventory Nursing Home Version (NPI) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Measures neuropsychiatric symptoms outcomes and caregiver burden - completed by primary caregiver
Clinical Global Impression Scale: Severity (CGI-S) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Indicates severity of dementia with agitation/aggression at the time of assessment - completed by physician
Mini Mental Status Examination (MMSE) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Measures cognition - primary caregiver completes with subject
Wechsler Adult Intelligence Scale 4th Edition (WAIS-IV) Digit Span (forwards and backwards) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Measures concentration, attention and memory - primary caregiver completes with subject
Geriatric Evaluation of Mental Status (GEMS) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Measures list learning tasks to assess verbal memory outcome - primary caregiver completes with subject
Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Measures functional ability outcomes - completed by primary caregiver
Use of Psychoactive "As Needed" (PRN) Medication | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Records use of PRN medication for agitation/aggression
Delirium and/or adverse reactions to ECT or medication | Participants will be followed on the average of 5 weeks (+/- 1 week) since ECT treatment is generally administered 3x per week for 4 weeks
  Assessed by treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Jack Mahdasian, MD, Principal Investigator — Pine Rest Christian Mental Health Services; Brent P Forester, MD, Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Older Adult Unit of Pine Rest Christian Mental Health Services, Grand Rapids, Michigan

REFERENCES:
- [Result] Ujkaj M, Davidoff DA, Seiner SJ, Ellison JM, Harper DG, Forester BP. Safety and efficacy of electroconvulsive therapy for the treatment of agitation and aggression in patients with dementia. Am J Geriatr Psychiatry. 2012 Jan;20(1):61-72. doi: 10.1097/JGP.0b013e3182051bbc. PMID 22143072